CLINICAL TRIAL: NCT04291339
Title: Comparison of the Efficacy of High-flow Nasal Oxygen Therapy and Facial Mask Ventilation on the Increase of the Oxygen Reserve Index During Anesthetic Induction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2019-1336
Record Dates: First submitted 2020-02-28; First posted 2020-03-02 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Adult Patients 20 Years of Age or Older Who Are Planning to Undergo Surgery Under General Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-flow nasal oxygen technique (Experimental): High-flow nasal oxygen will be applied to the patients through nasal openings using Optiflow system during anesthetic induction. Pulse oximetry and oxygen reserve index will be monitored continuously.
  Interventions: Procedure: High-flow nasal oxygen technique
- Mask ventilation technique (Active Comparator): Oxygen will be supplied through the mouth and nose to the patients using facial mask during anesthetic induction. Pulse oximetry and oxygen reserve index will be monitored continuously.
  Interventions: Procedure: Mask ventilation technique

INTERVENTIONS:
Procedure: High-flow nasal oxygen technique — High-flow nasal oxygen will be applied to the patients through nasal openings using Optiflow system during anesthetic induction. Pulse oximetry and oxygen reserve index will be monitored continuously.
  Arms: High-flow nasal oxygen technique
Procedure: Mask ventilation technique — Oxygen will be supplied through the mouth and nose to the patients using facial mask during anesthetic induction. Pulse oximetry and oxygen reserve index will be monitored continuously.
  Arms: Mask ventilation technique

SUMMARY:
The purpose of this study is to compare the ability of oxygenation with high-flow nasal oxygen therapy and mask ventilation technique for induction of anesthesia in adult patients who are planning to undergo surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged over 19 years who are scheduled for sleep endoscopy

Exclusion Criteria:

* basal skull fracture
* facial anomaly
* consciousness disorder
* Risk of aspiration
* necessity of awake fiberoptic intubation due to the large vocal cord mass, endotracheal tumor or bleeding.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-01-12 (Actual)

PRIMARY OUTCOMES:
Peak oxygen reserve index value | for 10 minutes during anesthetic induction. At Day 0.
  Oxygen reserve index will be monitored continuously during anesthetic induction.

SECONDARY OUTCOMES:
The time to achieve the peak oxygen reserve index value | for 10 minutes during anesthetic induction. At Day 0.
  Oxygen reserve index will be monitored continuously during anesthetic induction.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park S, Kim SY, Kim MS, Park WK, Byon HJ, Kim HJ. Comparison of preoxygenation efficiency measured by the oxygen reserve index between high-flow nasal oxygenation and facemask ventilation: a randomised controlled trial. BMC Anesthesiol. 2023 May 9;23(1):159. doi: 10.1186/s12871-023-02126-9. PMID 37161369